CLINICAL TRIAL: NCT04729933
Title: Implantation of a Permanent Interatrial Shunt to Reduce Left Atrial Filling Pressures Following MitraClip: The V-Wave Shunt MitraClip Study
Brief Title: Implantation of a Permanent Interatrial Shunt to Reduce Left Atrial Filling Pressures Following MitraClip
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: samir kapadia (Other)
Collaborators: V-Wave Ltd (Industry)
Responsible Party: Sponsor-Investigator, samir kapadia, Sponsor/Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200329; IRB 21-068 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Mitral Regurgitation
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): V-Wave Shunt Placement
  Interventions: Device: V-Wave Shunt Placement

INTERVENTIONS:
Device: V-Wave Shunt Placement — After the MitraClip Placement and after final screening, the existing transseptal puncture used for MitraClip placement is used to place the V-WAVE Shunt device.

SUMMARY:
This is an investigator initiated, prospective study to demonstrate the safety and feasibility of implantation of the V-Wave Interatrial Shunt System (herein called the "V-Wave Shunt" in patients immediately following percutaneous mitral valve repair using the MitraClip system.

DETAILED DESCRIPTION:
The V-Wave Shunt is a device placed across the interatrial septum (IAS) by cardiac catheterization which allows for the transfer of blood from the left atrium (LA) to right atrium (RA). The intended effect is to reduce excessive left-sided cardiac filling pressures in patients with advanced heart failure (HF) and thus improve symptoms related to pulmonary congestion. All patients in the study must meet all anatomic and clinical eligibility in the FDA approved indications for use of the MitraClip in functional mitral regurgitation (MR). All patients must have persistence of New York Heart Association (NYHA) class III or ambulatory class IV HF symptoms despite maximally tolerated guideline directed medical therapy (GDMT) as assessed by a Cardiologist specialist in advanced heart failure (HF). All patients will have reduced left ventricular (LV) ejection fraction (EF) ≥ 20% and ≤ 50% and at least moderate to severe 3-4+ MR with a functional or combined functional and degenerative mechanism. Despite MitraClip treatment and maximum GDMT, these patients are at high risk for recurrent HF events and readmission, and thus there is an unmet need for further therapies to improve outcomes in this patient population.

The existing transseptal puncture used for MitraClip placement will be used to place the V-Wave Shunt device after MitraClip placement.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must meet clinical and anatomic eligibility for commercial placement of MitraClip for functional MR, as specified by the MitraClip Instructions for Use (IFU).

a. Clinical eligibility for MitraClip: i. Symptomatic secondary MR (moderate-severe [3+ or 4+] or greater) due to ischemic or non-ischemic cardiomyopathy ii. NYHA functional class III, or ambulatory IV iii. Maximization of GDMT as directed by the "Heart Team", including an interventional cardiologist (implanting physician), heart failure cardiologist, and cardiothoracic surgeon. This includes adequate treatment for systolic HF (LV dysfunction), rhythm disorders, and coronary disease, if applicable

1. An inhibitor of the reninangiotensin system (RAS inhibitor), including an angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) or angiotensin receptor-neprilysin inhibitor (ARNI) and a beta-blocker (BB)
2. Other medications recommended for selected populations, e.g., mineralocorticoid receptor antagonist (MRA) or nitrates/hydralazine should be used in appropriate patients, according to the published guidelines.
3. Patient has been on stable HF medications as determined by the investigator, for at least 1 month, with the exception of diuretic therapy. Stable is defined as no more than a 100% increase or 50% decrease in dose within these periods.
4. Drug intolerance, contraindications, or lack of indications must be attested to by the investigator.
5. Receiving Class I recommended cardiac rhythm management device therapy.

   1. If indicated by class I guidelines, cardiac resynchronization therapy (CRT), implanted cardioverter-defibrillator (ICD) or a pacemaker should be implanted at least 3 months prior to device implantation
   2. These criteria may be waived if a patient is clinically contraindicated for these therapies or refuses them and must be attested to by the investigator.

iv. At least one hospitalization for heart failure in last year OR corrected BNP ≥ 300 pg/mL or corrected NTproBNP ≥ 1500 pg/mL v. Heart team has determined that mitral valve (MV) surgery will not be offered as a treatment option b. Anatomic eligibility for MitraClip: i. LVEF ≥ 20% and ≤ 50% ii. LV end-systolic dimension ≤ 70 mm iii. MV orifice area > 4.0 cm2 by TEE iv. Minimal calcification in the grasping area v. No leaflet cleft in the grasping area vi. In patients with a degenerative component to MR, the following additional criteria must be met:

1. Flail width <15 mm
2. Flail gap <10 mm vii. The primary regurgitant jet is non-commissural, and in the opinion of the implanting investigator can be successfully be treated by the MitraClip (if a secondary jet exists, it must be considered clinically insignificant) viii. Transseptal catheterization and femoral vein access is feasible per investigator 2. Provide written informed consent for study participation and be willing and able to comply with the required tests, treatment instructions and follow-up visits.

Exclusion Criteria:

Preliminary Exclusion Criteria (PEC) - to assessed by the Preliminary Screen at the baseline visit:

1. Severe pulmonary hypertension, defined as RV systolic pressure or PA systolic pressure > 70 mmHg, or PVR > 4 Woods units, measured by any modality (TTE, TEE, cardiac MRI, or pulmonary artery catheterization [if data available]).
2. Moderate or severe RV dysfunction defined as TAPSE <12mm or RVFAC ≤25% as assessed on Baseline TTE, or qualitative assessment of severe RV dysfunction on TTE, TEE, or cardiac MRI.
3. Untreated severe (3+ to 4+) tricuspid or pulmonary regurgitation.
4. Untreated clinically significant coronary disease requiring revascularization
5. Coronary artery bypass grafting, percutaneous coronary intervention, transcatheter aortic valve implantation, or CRT-D implantation within 30 days
6. Aortic or tricuspid valve requiring surgery or transcatheter intervention
7. COPD requiring continuous home oxygen therapy or chronic outpatient steroid use
8. Cerebrovascular accident within prior 30 days
9. Known severe symptomatic carotid stenosis
10. Carotid surgery or stenting within prior 30 days
11. ACC/AHA Stage D heart failure
12. Presence of any of the following:

    1. Hypertrophy cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
    2. Infiltrative cardiomyopathy (e.g. amyloidosis, hemochromatosis, sarcoidosis)
13. Leaflet anatomy which may preclude MitraClip implantation
14. Hemodynamic instability defined as systolic pressure < 90 mmHg with or without afterload reduction, cardiogenic shock or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device.
15. Need for surgery within 12 months
16. Life expectancy < 1 year due to non-cardiac conditions
17. Status 1 for cardiac transplant or history of cardiac transplant
18. Modified Rankin score ≥ 4 for disability
19. Prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure
20. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
21. Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (i.e., noncompliant, perforated)
22. Active infection requiring antibiotic therapy
23. TEE is contraindicated or high risk
24. Pregnant or planning pregnancy within 12 months
25. Known hypersensitivity or contraindication to procedural medications that cannot be adequately treated
26. Known allergy to nickel.
27. Patient is otherwise not appropriate for the study as determined by the investigator or the Eligibility Committee, for which the reasons must be documented.
28. Patient belongs to a vulnerable population per investigator's judgment or patient has any kind of disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures.

    Final Exclusion Criteria (FEC) - Assessed by the Final Screening, performed at time of cardiac catheterization prior to device placement (Study Intervention Visit)
29. Presence of severe pulmonary hypertension assessed by invasive hemodynamic measurement with pulmonary artery catheterization prior to MitraClip placement, defined as PA systolic pressure > 70 mmHg or PVR > 4 Woods units.
30. Anatomical anomaly on TEE that precludes implantation of the study device across the interatrial communication created by the MitraClip procedure, including:

    1. A posterior rim between the septum secundum and aorta (i.e. aortic rim) of < 5 mm.
    2. Atrial septal aneurysm defined as ≥ 10 mm of phasic septal excursion into either atrium or a sum total excursion of ≥ 15 mm during the cardiorespiratory cycle, with a base of ≥ 15 mm.
31. Moderate or worse MR ≥2+ at the end of MitraClip treatment (i.e. MR must be <2+ by TTE, TEE, invasive hemodynamics, or left ventriculography)
32. Key hemodynamic exclusions after MitraClip treatment:

    1. Mean LAP ≤ 20 mmHg following final result from MitraClip placement (i.e. mean LAP must be elevated > 20 mmHg after completion of MitraClip).
    2. Difference between mean LAP and mean RAP < 5mmHg after MitraClip placement (i.e. difference between LAP - RAP must be ≥ 5 mmHg).
    3. If the patient meets these hemodynamic exclusion criteria and mean arterial pressure (MAP) is < 90 mmHg, the MAP may be increased to ≥ 90 mmHg and repeat pressure measurements obtained in order to evaluate eligibility.

    i. IV fluids and medications may be given to support MAP to a goal ≥ 90 mmHg if necessary.
33. Characteristics of septal defect

    1. Angle of placement of V-WAVE shunt should be no more than 135 degrees to prevent slippage through the septum, and
    2. Septal defect created by MtrraClip delivery system must be 8mm or smaller, in any dimention, without evidence of a tear in the septum
34. Patient is otherwise not appropriate for study as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | Up to 1 month post implant
  Number of death caused by any condition
Stroke/paradoxical embolism | Up to 1 month post implant
  Number of patients who developed stroke/paradoxical embolism
Myocardial infarction | Up to 1 month
  Number of patients who developed MI
V-Wave shunt device embolization | Up to 1 month
  Number of V-Wave shunt device embolization occurrence
Cardiac Tamponade | Up to 1 month
  Number of occurrence of cardiac tamponade
Device related re-intervention or surgery | Up to 1 month
  Occurrence of device related re-intervention of surgery

SECONDARY OUTCOMES:
All-cause death | At 6 months, 1 year, 2 years, 3 years and 5 years
  Number of death caused by any condition
Stroke/paradoxical embolism | At 6 months, 1 year, 2 years, 3 years and 5 years
  Number of patients who developed stroke/paradoxical embolism
Myocardial infarction | At 6 months, 1 year, 2 years, 3 years and 5 years
  Number of patients who developed MI
V-Wave shunt device embolization | At 6 months, 1 year, 2 years, 3 years and 5 years
  Number of V-Wave shunt device embolization occurrence
Cardiac Tamponade | At 6 months, 1 year, 2 years, 3 years and 5 years
  Number of occurrence of cardiac tamponade
Device related re-intervention or surgery | At 6 months, 1 year, 2 years, 3 years and 5 years
  Occurrence of device related re-intervention of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kapadia, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No